CLINICAL TRIAL: NCT01960556
Title: Simulation-Based Pediatric Intensive Care Unit Central Venous Line Maintenance Bundle Education
Brief Title: Simulation-Based Central Venous Line Maintenance Bundle Education
Acronym: CA-BSI
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kiran Hebbar, Medical Director, Pediatric Simulation Center, Children's Healthcare of Atlanta
Other Study IDs: CA-BSI and Simulation
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Central Line Infection
Keywords: simulation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Simulation: Simulation Training part of education
  Interventions: Other: Simulation Training
- Non-Simulation Based Education: Did not receive simulation based education

INTERVENTIONS:
Other: Simulation Training — Simulation training provided to one group
  Other Names: Education
  Groups: Simulation

SUMMARY:
Catheter associated blood stream infections (CA-BSI) remain a source of significant morbidity and mortality in adult and pediatric critical care units. While it has been established that CVL maintenance bundles are pivotal to achieving and maintaining low CA-BSI rates, training and retention of proper bundle compliance remains a challenge.

The investigators prospectively compared this simulation-based program to a standard educational approach.

The investigators hypothesized that implementation of bedside simulation-based training of CVL dressing changes by registered nurses would improve CVL maintenance bundle compliance.

DETAILED DESCRIPTION:
The 2006 NACHRI Quality Transformation Effort demonstrated that additional reduction in pediatric catheter associated blood stream infection (CA-BSI) rates could be achieved through improving compliance with maintenance bundle care for central lines. The investigators objective was to improve maintenance bundle compliance rates and nursing competency surrounding central venous line (CVL) care in their pediatric intensive care unit (PICU).

A multidisciplinary team developed a bedside simulation-based training program to improve compliance with standard PICU CVL maintenance bundle. The investigators then performed a randomized comparison study comparing a standard CVL bundle education process for bedside PICU nurses in a control group (CG) to an intervention group (IG) receiving bedside training to simulate a CVL dressing change and maintenance bundle followed by intermittent educational refresh. Groups were assessed for compliance with prescribed components of the CVL bundle maintenance (CVL score).

CVL scores will be compared between groups

ELIGIBILITY:
Inclusion Criteria:

* Any nurse assigned to the PICU on a regular basis was eligible to participate in the study, including full-time, part-time, and occasional (prn) PICU nursing staff, as well as central staffing office (ICU float nurses) and traveler nurses contracted to the PICU for a minimum of 12 weeks

Exclusion Criteria:

* Nurses floating from other units, agency nursing personnel, or traveler nurse contract of < 12 week period were excluded. Nurses on orientation were excluded until completion of introductory 6-month probation period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric ICU nurses
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
CVL scores | 12 months
  Change in CVL scores with and without simulation based education

CONTACTS AND LOCATIONS:
Overall Officials: Kiran B Hebbar, MD, Principal Investigator — Children's Healthcare of Atlanta

REFERENCES:
- [Derived] Hebbar KB, Cunningham C, McCracken C, Kamat P, Fortenberry JD. Simulation-based paediatric intensive care unit central venous line maintenance bundle training. Intensive Crit Care Nurs. 2015 Feb;31(1):44-50. doi: 10.1016/j.iccn.2014.10.003. Epub 2014 Nov 22. PMID 25468293